CLINICAL TRIAL: NCT04619784
Title: The Effect of Pilates Application on Abdominal Muscle Function, Core Stability, Musculoskeletal Pain, Quality of Life, Anxiety and Depression in Parkinson's Patients
Brief Title: Effect of Pilates Application on Abdominal Muscle Function, Core Stability, Musculoskeletal Pain, Quality of Life, Anxiety and Depression in Parkinson's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Evrim Goz, Research assistant, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DokuzEU2
Record Dates: First submitted 2020-08-04; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease; Pilates; Muscle Function
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Demographic features will be questioned and recorded in the data recording form through face to face interview in patients who meet the inclusion criteria; evaluations will be made regarding muscle thickness and pain. Patients will receive 12 sessions of pilates. Patients will be evaluated before treatment, after treatment, at the 3rd and 6th months.
  Interventions: Other: Pilates Exercises
- Control Group (Other): Demographic features will be questioned and recorded in the data recording form through face to face interview in patients who meet the inclusion criteria; evaluations will be made regarding muscle thickness and pain. Their routine medical treatments were continued
  Interventions: Other: control

INTERVENTIONS:
Other: Pilates Exercises — Patients will receive 12 sessions of pilates.
  Arms: Treatment Group
Other: control — Their routine medical treatments were continued
  Arms: Control Group

SUMMARY:
In this study, it is aimed to investigate the effect of Pilates application on abdominal muscle function, core stability, musculoskeletal pain, quality of life, anxiety and depression in Parkinson's Patients.

DETAILED DESCRIPTION:
Objective: In this study, it is aimed to investigate the effect of Pilates application on abdominal muscle function, core stability, musculoskeletal pain, quality of life, anxiety and depression in Parkinson's Patients.

Method: The study included 15 Idiopathic Parkinson's Patients over 18 years of age, under stage 3 according to the Hoehn-Yahr clinical staging. Patients were divided into intervention and control groups. Pilates training was performed for 6 weeks, twice a week and 60 minutes per session in intervention group. Demographic features will be questioned and recorded in the data recording form through mutual interview in patients who meet the inclusion criteria; evaluations will be made regarding muscle thickness and pain. All patients will be evaluated before treatment, after treatment, at the 3rd and 6th months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Idiopathic Parkinson's Disease
* Must be older 18 years old
* Must have 24 and above score on Mini Mental Test
* Must be the third or lower stage according to the Hoehn-Yahr staging
* Must have stable clinical status

Exclusion Criteria:

* Musculoskeletal or cognitive impairment at a level affecting evaluation and treatment
* Other neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Function | Patients will be evaluated before treatment, 1 week after treatment, at the 3rd and 6th months after treatment
  Muscle thickness measurement will be used to evaluate the function of transversus. Ultrasonography with a linear transducer (MHz) will use to measure the Transversus Abdominis thickness both at rest and during the abdominal drawing-in maneuver (ADIM). During ADIM, participants will be asked to abdominal hollowing which will be a gentle voluntary contraction of abdominal wall. All images are obtained at the end of expiration not to allow the effect of respiration on muscle thickness. Three measures are recorded in the both condition. The average values of measures are used in the data analysis.

SECONDARY OUTCOMES:
Core stability | Patients will be evaluated before treatment, 1 week after treatment, at the 3rd and 6th months after treatment
  "Core" endurance and "core" power are the specific components of "core" stability and will be evaluated separately.
Musculoskeletal Pain | Patients will be evaluated before treatment, 1 week after treatment, at the 3rd and 6th months after treatment
  Musculoskeletal pain will be evaluated with The Nordic Musculoskeletal Questionnaire. Questionnaire includes 27 items exploring the presence of musculoskeletal symptoms during a 12-month period covering in nine different parts of the body (i.e. neck, shoulders, elbows, wrists/hands, upper back, lower back, hips/tights, knees, ankles/feet) [21]. It also has items pertaining to severity grades, determined according to functional status and the presence of musculoskeletal symptoms during the last seven days. All answers are given according to a dichotomous 'yes/no' response.The Turkish version of the NMQ has appropriate psychometric properties, including good test-retest reliability, internal consistency and construct validity.
Quality of Life | Patients will be evaluated before treatment, 1 week after treatment, at the 3rd and 6th months after treatment
  Quality of Life will be evaluated with 8-Item Parkinson's Disease Questionnaire / PDQ-8.The PDQ-8 is a brief form of the PDQ-39. One question from each of the eight domains on the PDQ-39 which are activities of daily living, bodily discomfort, cognition, communication, emotional well-being, mobility, social support, and stigma was chosen based on the strength of its correlation with the total domain score. Each question was scored from 0-4 points, and the scores were summed. The summed score was then divided by total possible score, and given as a percentage score out of 100.
Anxiety | Patients will be evaluated before treatment, 1 week after treatment, at the 3rd and 6th months after treatment
  Anxiety will be evaluated with Beck Anxiety Inventory. It is a 21-item questionnaire that includes 4-point Likert-type options with a score of 0-3 and measures the level of anxiety. The higher the total score indicates the severity of anxiety.
Pain intensity | Patients will be evaluated before treatment, 1 week after treatment, at the 3rd and 6th months after treatment
  Pain intensity will be evaluated with Visual Analog Scale. 10 cm long horizontal or vertical, numbered 1-10 forms are used.0 means no pain, 10 means unbearable pain.
Depression | Patients will be evaluated before treatment, 1 week after treatment, at the 3rd and 6th months after treatment.
  Depression will be evaluated with Beck Depression Inventory. It is a 21-item scale. The items contain sentences of four degrees that progress from less to more, which the participant will evaluate himself. The scale can be scored between 0 and 63. The high total score indicates the severity of the depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No